CLINICAL TRIAL: NCT04529993
Title: An Atlas of Airways at a Single Cell Level in Chronic Obstructive Pulmonary Disease, Idiopathic Pulmonary Fibrosis and Controls
Acronym: DISCOVAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-PP-06
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Interstitial Pulmonary Fibrosis
Keywords: lung; nasal mucosa; respiratory mucosa
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interstitial pulmonary fibrosis (Experimental)
  Interventions: Procedure: Bronchoscopy
- Chronic obstructive pulmonary disease (Experimental)
  Interventions: Procedure: Bronchoscopy
- Healthy volunteers (Experimental)
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Multiple level sampling of the respiratory mucosa (cytology brush and biopsies forceps)

SUMMARY:
The increasing incidence of chronic respiratory disease is a public health problem that affects hundreds of thousands of people worldwide at all ages. Directly exposed to atmospheric airborne contaminants (pollution, allergens), the respiratory tract represents a complex ecosystem involving different cells (multiciliated, basal, mucosecretory, neuroendocrine, etc.) that develop complex interactions with the surrounding connective tissue but also with their rich immune environment and the local microbiota. Although a pathophysiological continuum is postulated between the nasal and bronchial airways in certain diseases, such as allergic diseases, investigators have demonstrated large gene expression gradients between samples taken from the nasal and bronchial airways in different studies. Specifying the cellular variability throughout the respiratory tree in a normal physiological situation is one of the major objectives defined in the establishment of an atlas of all airway cells, as defined in the objectives of the international consortium Human Cell Atlas.

The sequencing of the RNAs present specifically in each individual cell ("single-cell RNAseq"), and its comparison with neighbouring cells allows to document the precise cellular contributions, as well as the signalling pathways involved. The development of tissue sampling, stabilization, transport and single cell analysis procedures can be performed on primary respiratory epithelium cultures and can also be extended to respiratory samples from healthy volunteers.

This project will analyze gene expression profiles at the single cell level (single cell RNAseq) in volunteers with chronic obstructive pulmonary disease, interstitial pulmonary fibrosis and compared to healthy subjects of the same age. The technical modalities of the samples will be brushing and staged airway biopsies for direct analysis of the samples. This approach will be complemented by an air-liquid interface culture to allow secondary analysis in single cell RNAseq and three-dimensional mapping of the distribution of these cells with single cell in situ analysis.

Thanks to sampling at several levels of the respiratory tree (nose, bronchioles, bronchioles), cellular and gene expression variations along the tracheobronchial axis will be exhaustively documented in subjects of different ages, healthy or suffering from pathologies such as chronic obstructive pulmonary disease and interstitial pulmonary fibrosis. These data will serve as worldwide references for comparisons in different physiological and pathological contexts.

ELIGIBILITY:
Inclusion Criteria:

* Absence of acute pathology
* Absence of symptom evoking an evolutionary pathology

For healthy volunteers :

* Non-smoker (active or passive) or ex-smoker of less than 5 packet-years and quit for more than 10 years.
* Absence of known significant chronic pathology
* Normal Respiratory Function Test (RFT)
* Woman of childbearing age using an effective method of contraception

For COPD patients :

* Diagnosis of COPD based on dyspnea, chronic cough or sputum production, a history of recurrent lower respiratory tract infections and/or a history of exposure to risk factors for the disease associated with spirometry that demonstrates a post-bronchodilator FEV1/FVC ratio < 0.70 and lack of reversibility.
* Stage GOLD 1 (post-bronchodilator FEV1 ≥ 80% theoretical) or 2 (post-bronchodilator FEV1 between 50 and less than 80% theoretical) or 3 (post-bronchodilator FEV1 between 30 and less than 50% theoretical) For IPF patients
* Diagnosis of idiopathic pulmonary fibrosis made less than 5 years ago on the basis of scannographic and/or histological criteria and validated at a consultation meeting on interstitial pathology according to the ATS/ERS/JRS/ALAT 2018 recommendations.

Exclusion Criteria:

* Recent rhino-bronchial infection (< 6 weeks)
* Subjects on antiplatelet or other anticoagulant medication at risk of bleeding during sampling.
* Subjects with a history of clinically significant vaginal discomfort (i.e., recurrent or unconsciousness, etc.)
* History of allergy or intolerance to xylocaine and/or propofol
* History of significant epistaxis (i.e. recurrent epistaxis of any quantity or at least one severe epistaxis)
* Subject at risk of difficult intubation according to the criteria of the 2006 FSSR expert conference*.
* Pregnant (a urine test will be performed for all women of childbearing age) or breastfeeding woman

For patients :

* Long-term systemic corticosteroid therapy regardless of the reason for the prescription.
* Systemic corticosteroid therapy within the previous 3 months
* Patient on long-term oxygen therapy
* Chronic cardiovascular, neuro-psychic, metabolic pathology in progress, clinically significant or uncontrolled in the last 6 months
* Other associated chronic respiratory pathology (COPD, asbestosis, bronchiectasis ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Number of samples usable | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie LEROY, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No